CLINICAL TRIAL: NCT00219830
Title: Health and Social Inequalities in the Uptake of Cardiac Rehabilitation in Northern Ireland: an Alternative Program for Non-attenders: (2) a Randomised Controlled Trial.
Brief Title: A Trial of a Home Based Walking Program as an Alternate Program for Non Attenders at Cardiac Rehabilitation
Acronym: CRU-SHAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no invited participants agreed to undertake the proposed intervention
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Dr Margaret E Cupples, Professor, Queen's University, Belfast
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COM2376-02-02
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Acute Myocardial Infarction
Keywords: Cardiac Rehabilitation; Walking; Acute Myocardial Infarction; Secondary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - home-based walking program (Experimental): Based on medical record held in general practice, patients who had not attended a formal cardiac rehabilitation program after myocardial infarction and were enrolled in home-based walking programme
  Interventions: Behavioral: home-based walking program
- 2 - cardiac rehabilitation (No Intervention): Based on medical record held in general practice, patients who are identified as having attended a Cardiac Rehabilitation program following myocardial infarction - 'usual care'

INTERVENTIONS:
Behavioral: home-based walking program — Home-based walking program; included use of pedometer and daily walk diary
  Arms: 1 - home-based walking program

SUMMARY:
The purpose of this study is to investigate if a home-based walking program is an acceptable alternative for those who choose not to attend formal cardiac rehabilitation programs and if such a program has an effect on coronary risk or physical fitness.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is the most important cause of life years lost in Northern Ireland (NI). A recently updated Cochrane review (Joliffe et al, 2003) confirmed the findings of earlier meta-analyses (O'Connor et al, 1989; Oldridge et al, 1988) which indicated that participation in cardiac rehabilitation (CR) reduces mortality after MI. The earlier work demonstrated a reduction of 20-25% in all-cause and cardiac mortality. The recent work allowed analysis of an increased number of patients (8440 in 32 trials) and reported a reduction in total cardiac mortality of up to 31%. Participation in CR after MI also improves well-being and reduces disability (NHS, 1998). However, informal reports suggest that only approximately 50% of patients actually attend a hospital based program.

The hypothesis to be tested is that for those who chose not to attend formal CR, a home-based walking program is an acceptable alternative.

This programme of work entails two separate study designs. To evaluate the home-based walking program, we plan a randomised controlled trial (RCT). Randomisation of subjects to study groups will follow determination of eligibility to participate. Participants randomised to the experimental group will be asked to walk for up to 30 minutes, 5-days per week. They will be requested to record aspects of their walking in a diary, including time, intensity and number of steps taken (recorded using a pedometer).

Qualitative methodology using semi-structured interviews will be used to explore the experiences of those allocated to the intervention group. The attitudes and experiences of other non-attenders of CR who declined to participate in the trial will be explored in focus groups. Three focus groups each containing 8 participants are planned.

Focus group transcripts will be analysed independently by two observers using a computer program (NUDIST) to identify themes and develop questions for the semi-structured interviews. Analysis of the semi-structured interviews will be descriptive, responses being categorised into themes as appropriate.

RCT results will be analysed by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Justification of diagnosis of myocardial infarction by report of cardiac bio-markers or electrocardiogram changes

Exclusion Criteria - planned for RCT - applied to small pilot:

* Heart failure/ Cardiogenic shock
* Complex ventricular arrhythmias
* Mental/physical impairment (exclude if housebound/dementia)
* Valve disorder-severe stenotic or regurgitant lesion
* Hypertrophic cardiomyopathy
* Exercise Stress Test result- exclude if ST depression>=2 mm or angina at <5 Metabolic Equivalent of Tasks (METS) (e.g. 3 minutes of a Bruce protocol). (Also exclude if report of ST segment depression >=1 mm on resting ECG )

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-01 (Estimated); Primary Completion 2007-05 (Estimated); Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Score | 16-20 weeks post myocardial infarction
  MacNew Post-myocardial infarction questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E Cupples, MD, Principal Investigator — Queen's University, Belfast; Mark A Tully, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Dept of General Practice, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data - these will form an aggregated database for determination of the design of a later definitive study.

REFERENCES:
- [Background] Tully M, Cupples ME, Young IS et al. CRU-SHAL Study - provision and uptake of cardiac rehabilitation in Northern Ireland. British Association for Cardiac Rehabilitation Annual Conference: Emerging Challenges for Cardiac Rehabilitation. September 2006, p10.